CLINICAL TRIAL: NCT02615717
Title: Using Attentional Bias Modification to Address Trauma Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Responsible Party: Principal Investigator, Christina Hein, Clinical Psychology Graduate Student, University of Nebraska Lincoln
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNebraskaLincoln
Record Dates: First submitted 2015-11-23; First posted 2015-11-26 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-12

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attentional Bias Modification (Experimental): In the ABM treatment condition, participants will have four 20-minute in-lab treatment conditions across two weeks. Within these Attention Bias Modification sessions, participants will be presented with a fixation cross for 500 ms. The fixation cross will then be replaced with a word pair consisting of either a threat/neutral pair or a neutral/neutral word for 500 ms, followed by a probe in the location of one of the two words (80% threat/neutral pairs, 20% neutral/neutral pairs; the target will always appear in the location of the neutral word).
  Interventions: Behavioral: Attention Bias Modification
- Attentional Control Condition (Active Comparator): Participants will have four 20-minute in-lab treatment conditions across two weeks. Within the Attention Bias Modification control sessions, participants will be presented with a fixation cross for 500 ms. The fixation cross will then be replaced with a word pair consisting of either a threat/neutral pair or a neutral/neutral word for 500 ms, followed by a probe in the location of one of the two words (80% threat/neutral pairs, 20% neutral/neutral pairs; the target appears in the location of the neutral word in 50% of the trials. Complete Stroop and 3-back task, etc.
  Interventions: Behavioral: Attention Bias Modification

INTERVENTIONS:
Behavioral: Attention Bias Modification — comparison of treatment versus control

SUMMARY:
Threat-related attentional biases have been identified as a possible precursor to the onset and maintenance of posttraumatic stress disorder (PTSD). As a result, protocols such as Attention Bias Modification (ABM) have been developed and utilized to treat these attentional biases in adults diagnosed with PTSD. However, to-date, ABM protocols have not been examined for use specifically among victims of sexual assaults. Participants are 20 undergraduate women enrolled in a Midwest university. The efficacy of ABM in this population will be assessed, as will the relationship between ABM and PTSD symptom clusters and outcome variables such as anxiety and depression scores.

DETAILED DESCRIPTION:
A relatively new intervention designed to reduce attention toward (or minimize disengagement from) threat-related information is attention bias modification (ABM). ABM is a novel treatment that may address several limitations posed by the use of CPT and PE. ABM is typically administered via computer, involving brief 20-minute sessions in which participants are trained to disengage from the threat cues to which they are naturally attuned. ABM addresses attentional biases in a similar, though more direct, manner as does CBT through the use of uninterrupted, repetitive exposure to feared threat cues or words in order to allow the patient to interpret that feared objects and situations are safe. In particular, ABM's effectiveness arises through the intent to normalize both attentional biases towards and away from threats such that the intended outcome is the non-existence of any bias surrounding threat cues. ABM addresses the specific bias in attention through targeting implicit, sub-cortical processes that focus on perturbed neural circuitry function. It trains individuals to remove any attention to or avoidance of threat cues by training brains to focus equally on threat and non-threat cues. Therefore, ABM further extends work implicating threat-related attention bias in anxiety disorders.

ABM has successfully improved or alleviated symptoms of many disorders, including anxiety disorders, depression, obsessive-compulsive disorder, and chronic pain. In addition, ABM has been successfully implemented in many populations such as inpatient active duty U.S. military members, Israeli Defense Force soldiers, pediatrics, and outpatients with chronic PTSD. Despite these findings, ABM has never been applied to individuals with current, lifetime, or chronic PTSD resulting from sexual assaults. Furthermore, studies assessing the use of ABM have found consistent benefits from ABM control groups, although this effect has been smaller than those in the ABM treatment groups. Authors contend that the reason that ABM control groups may have experienced a decrease in symptoms may be that the use of training (regardless of treatment or control status) improves the relationship between emotional stimuli and the response required by participants in order to learn to exert attentional control.

If ABM proves to be effective in addressing attentional biases associated with PTSD and its associated symptom clusters, it is a unique treatment that has the potential to address many of the limitations or concerns faced by those who rely exclusively on CPT or PE; benefits of ABM include that the treatment (1) is a relatively simple and brief intervention, (2) may be administered electronically and remotely at a patient's home or at locations beyond a typical clinical office, and (3) has the potential to be mass-administered. As ABM is a relatively new treatment with many implications for utilization, its full potential has not yet been explored; in particular, there are several ways with which ABM may interact with empirically supported treatments (ESTs) as CPT and PE.

Firstly, it is important to recognize that CPT and PE have both been criticized for their role in requiring participants to immediately "dwell in the past", frequently resulting in clients reporting distress. This is particularly true in individuals who may have potentially been coping with or managing their trauma reaction through the use of intense avoidance. Thus, as a prelude to integrating individuals into CPT or PE, ABM has the potential to be a useful transition prior to ESTs to increase tolerance and prepare individuals to transition and integrate into these more provocative types of treatments. Starting with a treatment such as ABM, which introduces individuals to non-specific trauma content, might serve to help people to be more amenable to other ESTs such as CPT or PE, ultimately increasing willingness to start and stay in therapy, decreasing attrition, and improving retention.

Secondly, ABM interventions have been shown in several populations to result in at least a mild reduction of symptoms. Even mild reductions of symptoms may open the door to allowing an individual to make larger improvements through more other evidence-based interventions. Studies show that individuals with more severe pretreatment trauma-related cognitions have slightly worse PE outcomes than do individuals beginning treatment with more moderate symptoms. In applying ABM prior to CPT or PE, it is likely that the mild reduction of symptoms beforehand may ultimately increase the effectiveness and efficiency of ESTs.

Current Study Despite recent focus on attention training in PTSD, researchers have not yet examined whether training procedures such as ABM are capable of modifying attentional biases in individuals whose most disturbing and impactful trauma is a sexual assault. Thus, in this current study, the investigators aimed to examine the effect of ABM in a sample of women who have previously experienced an adult sexual assault. The aims of this study are three-fold: first and foremost, as this is the first study of its kind to assess the efficacy of ABM treatment in a sample of sexual assault victims, the investigators will be examining the effect of ABM in reducing PTSD symptoms within this trauma type. Secondly, investigators are exploring what PTSD symptoms or symptom clusters predict treatment outcomes and attentional variability. Finally, investigators expect to quantify and document attention variability in this population, and will explore whether variability is predictive of treatment outcomes.

Regarding this study's aims, investigators hypothesize that (1) both the ABM treatment and control groups will experience decreased PTSD, depressive, and anxiety symptoms, but with a greater decrease from baseline in the treatment condition. Secondly, investigators hypothesize that (2) there will be a relationship between heightened symptom clusters as expressed by the individuals and their attentional biases, such that individuals high in avoidance symptoms (Criterion C on the Clinician-Administered PTSD Scale, CAPS-5) will demonstrate decreased response times to threat cues on measures of executive functioning with low variability, while those high in hyperarousal symptoms (Criterion E on the CAPS-5) will demonstrate increased response times and low variability. In contrast, investigators expect those high in both symptom clusters (hyperarousal and avoidance) will demonstrate high variability in reaction times, and those low in both symptom clusters will demonstrate low variability. Finally, investigators hypothesize that (3) increased attention variability will be associated with higher PTSD, depressive, and anxiety symptoms, but greater changes in attention variability across the study will be associated with greater improvements on PTSD, depressive, and anxiety symptoms. More specifically, investigators hypothesize that as a result of treatment, those participants who have the greatest decreases in variability over the course of treatment will be higher in hyperarousal and/or avoidance over those who are low in both symptom clusters.

ELIGIBILITY:
Inclusion Criteria:

* Female, 19+, have experienced at least one adult sexual trauma, and must currently be experiencing PTSD symptoms as a result of the sexual assault

Exclusion Criteria:

* male

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina L Hein, B.A., Principal Investigator — University of Nebraska Lincoln
Locations (1):
- University of Nebraska-Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aupperle RL, Melrose AJ, Stein MB, Paulus MP. Executive function and PTSD: disengaging from trauma. Neuropharmacology. 2012 Feb;62(2):686-94. doi: 10.1016/j.neuropharm.2011.02.008. Epub 2011 Feb 22. PMID 21349277
- [Background] Bar-Haim Y. Research review: Attention bias modification (ABM): a novel treatment for anxiety disorders. J Child Psychol Psychiatry. 2010 Aug;51(8):859-70. doi: 10.1111/j.1469-7610.2010.02251.x. Epub 2010 May 6. PMID 20456540
- [Background] Bar-Haim Y, Holoshitz Y, Eldar S, Frenkel TI, Muller D, Charney DS, Pine DS, Fox NA, Wald I. Life-threatening danger and suppression of attention bias to threat. Am J Psychiatry. 2010 Jun;167(6):694-8. doi: 10.1176/appi.ajp.2009.09070956. Epub 2010 Apr 15. PMID 20395400
- [Background] Carlbring P, Apelstrand M, Sehlin H, Amir N, Rousseau A, Hofmann SG, Andersson G. Internet-delivered attention bias modification training in individuals with social anxiety disorder--a double blind randomized controlled trial. BMC Psychiatry. 2012 Jun 25;12:66. doi: 10.1186/1471-244X-12-66. PMID 22731889
- [Background] Echiverri AM, Jaeger JJ, Chen JA, Moore SA, Zoellner LA. "Dwelling in the Past": The Role of Rumination in the Treatment of Posttraumatic Stress Disorder. Cogn Behav Pract. 2011 Aug;18(3):338-349. doi: 10.1016/j.cbpra.2010.05.008. PMID 22190846
- [Background] Eldar S, Apter A, Lotan D, Edgar KP, Naim R, Fox NA, Pine DS, Bar-Haim Y. Attention bias modification treatment for pediatric anxiety disorders: a randomized controlled trial. Am J Psychiatry. 2012 Feb;169(2):213-20. doi: 10.1176/appi.ajp.2011.11060886. PMID 22423353
- [Background] Hakamata Y, Lissek S, Bar-Haim Y, Britton JC, Fox NA, Leibenluft E, Ernst M, Pine DS. Attention bias modification treatment: a meta-analysis toward the establishment of novel treatment for anxiety. Biol Psychiatry. 2010 Dec 1;68(11):982-90. doi: 10.1016/j.biopsych.2010.07.021. PMID 20887977
- [Background] Iacoviello, B. M., Amir, N., Bar-Haim, Y., Beard, C., Montana, R., Kuckertz, J. W., … & De Raedt, R. (2014). Maximizing the effects of attention bias modification for anxiety: How and for whom. Symposium presented that the 48th annual congress presented at Associaion for Behavioral and Cognitive Therapies, 21 November 2014.
- [Background] Kuckertz JM, Amir N, Boffa JW, Warren CK, Rindt SE, Norman S, Ram V, Ziajko L, Webb-Murphy J, McLay R. The effectiveness of an attention bias modification program as an adjunctive treatment for Post-Traumatic Stress Disorder. Behav Res Ther. 2014 Dec;63:25-35. doi: 10.1016/j.brat.2014.09.002. Epub 2014 Sep 16. PMID 25277496
- [Background] Moser JS, Cahill SP, Foa EB. Evidence for poorer outcome in patients with severe negative trauma-related cognitions receiving prolonged exposure plus cognitive restructuring: implications for treatment matching in posttraumatic stress disorder. J Nerv Ment Dis. 2010 Jan;198(1):72-5. doi: 10.1097/NMD.0b013e3181c81fac. PMID 20061873
- [Background] Najmi S, Amir N. The effect of attention training on a behavioral test of contamination fears in individuals with subclinical obsessive-compulsive symptoms. J Abnorm Psychol. 2010 Feb;119(1):136-42. doi: 10.1037/a0017549. PMID 20141250
- [Background] Schoorl M, Putman P, Van Der Does W. Attentional bias modification in posttraumatic stress disorder: a randomized controlled trial. Psychother Psychosom. 2013;82(2):99-105. doi: 10.1159/000341920. Epub 2012 Dec 22. PMID 23295710
- [Background] Sharpe L, Ianiello M, Dear BF, Perry KN, Refshauge K, Nicholas MK. Is there a potential role for attention bias modification in pain patients? Results of 2 randomised, controlled trials. Pain. 2012 Mar;153(3):722-731. doi: 10.1016/j.pain.2011.12.014. Epub 2012 Jan 26. PMID 22281100
- [Background] Weathers, F. W., Blake, D. D., Schnurr, P. P., Marx, B. P., & Keane, T. M. (2013). The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). Interview available from the National Center for PTSD at www.ptsd.va.gov.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Attentional Bias Modification | Attentional Control Condition
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attentional Bias Modification | Attentional Control Condition | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.7 (1.2) | 21.7 (2.9) | 20.7 (2.2)
Gender [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Clinician-Administered PTSD Scale (CAPS-5)
Description: Assesses symptoms and severity of Posttraumatic Stress Disorder Range: 0-80; total score utilized. Higher values indicate higher severity Subscales are summed to create a total score; subscales made up of different facets of PTSD.
Time Frame: within three days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attentional Bias Modification | Attentional Control Condition
Number analyzed (Participants) | 3 | 3
units on a scale | 10.3 (10.2) | 10.0 (5.3)

2. Secondary Outcome: PTSD Checklist (PCL-5)
Description: Self-report of PTSD symptom severity Scale range: 0-80 Total score utilized, all items summed. Higher score indicates higher severity.
Time Frame: within three days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attentional Bias Modification | Attentional Control Condition
Number analyzed (Participants) | 3 | 3
units on a scale | 11.0 (8.2) | 10.0 (8.5)

3. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: Self-report measure of 9 symptoms related to depression Range: 0-27, all items summed Higher score indicates higher severity
Time Frame: within three days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attentional Bias Modification | Attentional Control Condition
Number analyzed (Participants) | 3 | 3
units on a scale | 5.3 (3.8) | 6.7 (4.5)

4. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: Self-report measure of 20 symptoms of anxiety Range: 0-60 all items summed Higher score indicates higher severity
Time Frame: within three days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attentional Bias Modification | Attentional Control Condition
Number analyzed (Participants) | 3 | 3
units on a scale | 29.0 (7.9) | 29.0 (6.0)

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events were not collected/assessed
Arm/Group | Attentional Bias Modification | Attentional Control Condition
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes